CLINICAL TRIAL: NCT06634342
Title: One-step HCV RNA Testing Among SSP Participants
Brief Title: One-step HCV RNA Testing Among SSP Participants (HOT Study)
Acronym: HOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Sara Glick, Associate Professor: Medicine- Allergy and Infectious Disease, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00021203
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Testing Effect of Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Participants of a syringe services program (Experimental): Participants of the syringe services program who will be offered point-of-care hepatitis C RNA testing will be adults 22 or older who do not already know they have HCV infection.
  Interventions: Diagnostic Test: HCV RNA Rapid testing

INTERVENTIONS:
Diagnostic Test: HCV RNA Rapid testing — Participants will receive point-of-care hepatitis C RNA testing using the GeneXpert IV Xpress System technology.

SUMMARY:
The HOT (HCV One-step Test) Study is an observational prospective study to evaluate the use of a recently FDA-approved point-of-care RNA test for hepatitis C virus (HCV) in a sample of clients of a syringe services program (SSP). We aim to answer the following questions:

1. How will point-of-care HCV RNA testing with Xpert, provided at an SSP, effect how people who use drugs receive their results, get linked to HCV care services, and initiate and complete HCV treatment> Aim 2: What are the most effective ways to implement point of care HCV RNA testing in syringe services programs?

DETAILED DESCRIPTION:
This study would be conducted in partnership with the Public Health - Seattle & King County SSP, which is the SSP that the project principal investigator is affiliated with in Seattle WA. The PHSKC SSP will be provided with a Cepheid Xpert HCV RNA machine and testing cartridges. Staff will be trained by Cepheid staff on the one-step HCV RNA testing protocol, including collecting blood from participants, using the test machine, interpreting results, and returning results to participants.

HCV testing and linkage to care activities will be monitored for six months as part of this study. Once all training and protocol development is complete, the PHSKC SSP will make the one-step HCV testing algorithm available to their clients and invite them to participate. SSP staff will conduct the one-step HCV testing and linkage algorithm according to the project protocol.

Clients who choose to be tested will participate in an informed consent process for study procedures. Participants who complete the HCV test and receive their results will receive a $15 incentive. All quantitative data related to the study will be entered directly into REDCap data collection tools. SSP staff who conduct testing will record a participant's HCV test result, whether/when they received their result, and whether/when they received a referral to HCV care. Participants will need to provide identifying information (e.g., name and birthdate) and sign a release of information form to facilitate longitudinal data collection on linkage to care and treatment initiation. SSP staff will use this information to follow up with providers to indicate whether/when participants attended an HCV care visit, whether/when participants began HCV treatment, and if they achieved cure (i.e., sustained viral response at 4 weeks). No other information will be requested or recorded from health care providers.

We will ask the PHSKC SSP to gather data on prior HCV testing and linkage efforts for the 6 months prior to the implementation of the one-step algorithm (standard of care). This will include any data that are available related to volume of HCV screening and RNA testing, participant receipt of results, and linkage to care efforts.

During the six months of the testing project, we will also conduct qualitative data collection. First, UW staff will conduct 12 in-depth interviews with participants who were involved in the testing component of the study. These interviews will be conducted with participants who received negative HCV RNA results, both those who were and were not linked to care, and those who started HCV treatment. The goal of these interviews will be to understand the participants' previous testing experiences and interest in HCV care, present testing experiences and interest in care, and overall impressions of the one-step testing algorithm. Staff will use purposive sampling to recruit participants and conduct private interviews using a semi-structured interview guide. Participants who complete these interviews will receive a $40 incentive.

Second, UW staff will conduct in-depth interviews with all staff at the PHSKC SSP who were involved with the HCV testing study to understand the experiences of staff who conducted the one-step testing algorithm compared to previous testing algorithms (e.g., HCV rapid screening and/or laboratory-based HCV RNA testing). Specific questions will assess facilitators and barriers to providing one-step HCV testing in SSPs, as well as recommendations for implementing similar protocols in other SSPs.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 22

Exclusion Criteria:

* Already knows they are infected with hepatitis C virus.
* past participation in this study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Receipt of HCV RNA test results | 6 months
  Percentage of individuals who complete a HCV RNA test and who also receive their test results.
Linkage to HCV care | 6 months
  Percentage of individuals who test positive for HCV who are connected with HCV treatment services
Cure rate | 6 months
  Percentage of individuals who are connected with HCV treatment who are cured of HCV.

SECONDARY OUTCOMES:
Testing willingness | 6 months
  Percentage of participants offered the HCV RNA test who agree to be tested
Testing results | 6 months
  Percentage of participants who receive an HCV RNA test who test positive for HCV

CONTACTS AND LOCATIONS:
Overall Officials: Sara Glick, PhD, MPH, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No